CLINICAL TRIAL: NCT02970461
Title: Gamifying Patient's Personal Data Validation and Completion in a Personal Health Record
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital Italiano de Buenos Aires (Other)
Collaborators: Salumedia Tecnologias (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2258
Record Dates: First submitted 2016-11-15; First posted 2016-11-22 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Chronic Disease
Keywords: personal health record; gamification; chronic patient care
MeSH Terms: conditions — Chronic Disease | interventions — Control Groups

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group (Placebo Comparator): Subjects will see in their Personal Health Record home page a simple text link pointing to their Bio page. Once in their Bio page, the site will display their personal information as usual with the only addition of a "validate data" button next to any non-validated field. The option to edit fields will also be present.
  Interventions: Other: Control Group
- Gamified Group (Experimental): Subjects will see in their Personal Health Record home page a graphical representation of the percentage of completeness their Bio page has that when clicked acts as a link to their Bio page. Once in their Bio page, the site will display graphical elements such grayed out fields, graphical representations of the percentage of completeness for each data group and on mouse hover over any field a tooltip will inform of what percentage of completeness will be awarded if the data is validated. Also, an addition of a "validate data" button next to any non-validated field. The option to edit fields will also be present.
  Interventions: Other: Gamified Group

INTERVENTIONS:
Other: Gamified Group — See Gamified Group in Arms description.
  Arms: Gamified Group
Other: Control Group — See Control Group in Arms description.
  Arms: Control Group

SUMMARY:
A randomized controlled trial design is used to test the efficacy of gamification elements to drive user behavior in a personal health record.

DETAILED DESCRIPTION:
Electronic personal health record systems (PHRs) support patient centered healthcare by making medical records and other relevant information accessible to patients, thus assisting patients in health self-management[1,2]. The Hospital Italiano de Buenos Aires (HIBA) is a private hospital in Buenos Aires, capital of Argentina. It has 500 beds and serves around 50,000 patients per month. Its main facilities cover a surface area of 78,000 m² (850,000 ft²). The hospital treats both private patients and those derived by social security. It also provides its own Health Maintenance Organization (HMO) being the most important pre-paid healthcare service in Argentina, with about 150,000 clients. HIBA has a Health Information System (HIS) and Electronic Health Records (EHR) since 1998 and implemented a PHR in 2007. The PHR gives patients access to aspects of the EHR related to their Health Care (laboratory, diagnosis, preventive information, medications lists), supports messaging with their physician, scheduling services and medication delivery for Self management, among other things. The majority of HIBA HMO affiliates are enrolled to this PHR. In 2015 HIBA underwent the process of accreditation by the United States Joint Commission[3]. As part of this process, HIBA redefined and refined the EHR/PHR data set, including new fields and regrouping pre-existent ones. EHR/PHR's personal data set is now composed of a series of fields grouped as depicted below. Personal data information is a difficult data set to capture, particularly those regarding social and cultural background information[4]. This data set is not only useful to help better healthcare system management, it is also relevant as it is used for epidemiological and preventive purposes[5-7].

Gamification is a term used to describe using game elements in non-game environments to enhance user experience[8,9]. It has been incorporated with commercial success into several platforms (Linkedin, Badgeville, Facebook). While over the past years gamification elements have been incorporated in healthcare scenarios there is still little evidence on how effective they are[10-12]. Game elements provide engagement consistent with various theories of motivation[13], positive psychology (e.g., flow)[14], and also provide instant feedback. Feedback is more effective when it provides sufficient and specific information for goal achievement and is presented relatively close in time to the event being evaluated. Feedback can reference individual progress, can make social comparisons, or can refer to task criteria.

In order to assess whether gamification is an effective tactic to drive PHR users' behavior, an intervention was designed. The investigators used gamification elements such as points, graphical representations and playful attitude to the design and interactions of the Bio page in the Hospital's PHR. These elements provide instant feedback to user actions. A control group with no game elements will be compared with a gamified group to see if these new game elements would increase patient's personal data rectification, validation and completion in the Hospital's PHR. A status variable was created and assigned to all fields according to the following scheme:

* Completed: user has modified empty field.
* Corrected: user has modified non-empty field.
* Verified: user has updated Group but field data has experienced no change.
* Validated: user has clicked on the "validate" button.

EHR/PHR Personal data set

1. Contact Information

   * First Name
   * Last Name
   * Date of Birth
   * ID Number
2. Nationality

   * Citizenship
   * Languages Spoken
3. Place of Residence

   * Street
   * Number
   * Floor
   * Zip Code
   * Town
   * Province
   * Country
4. E-Mail

   - E-mail address
5. Phone Numbers

   * Home Number
   * Work Number
   * Fax
6. Emergency Contact

   * First Name
   * Last Name
   * Relationship with patient
   * Address
   * Phone Number
7. Billing Information

   * Street
   * Number
   * Floor
   * Zip Code
   * Town
   * Province
   * Country
8. Social Aspects

   * Type of Residence
   * Living Situation
9. Education

   - Highest Academic Degree Achieved
10. Cultural Aspects

    - Religious Belief
11. Special Needs

ELIGIBILITY:
Inclusion Criteria:

* Patients enrolled in the Hospital Italiano de Buenos Aires system who are over 18 years old
* Patients who are registered in Hospital Italiano de Buenos Aires' Personal Health Record
* Patients whose use of the Personal Health Record during the previous year exceeds the median of use

Exclusion Criteria:

* Refusal to participate or to the informed consent process
* Subjects with a record of Obsessive Compulsive Disorders or related condition as per DSM IV
* Subjects with a record of Neurological conditions that could impair reading (aphasia, dementia, etc)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40000 (Estimated)
Dates: Start 2016-07; Primary Completion 2016-11 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Change in Number of Completed Fields | Measured at baseline, 30 days after and 6 months after
  See "Completed" and "EHR/PHR Personal data set" in Study Detailed Description for more information.

SECONDARY OUTCOMES:
Change in Number of Corrected Fields | Measured at baseline, 30 days after and 6 months after
  See "Corrected" and "EHR/PHR Personal data set" in Study Detailed Description for more information.
Change in Number of Validated Fields | Measured at baseline, 30 days after and 6 months after
  See "Validated" and "EHR/PHR Personal data set" in Study Detailed Description for more information.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Bonofiglio, MD, Study Chair — Hospital Italiano de Buenos Aires
Locations (1):
- Hospital Italiano de Buenos Aires, Gascon 450, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cahill JE, Gilbert MR, Armstrong TS. Personal health records as portal to the electronic medical record. J Neurooncol. 2014 Mar;117(1):1-6. doi: 10.1007/s11060-013-1333-x. Epub 2014 Jan 30. PMID 24477621
- [Background] Tang PC, Ash JS, Bates DW, Overhage JM, Sands DZ. Personal health records: definitions, benefits, and strategies for overcoming barriers to adoption. J Am Med Inform Assoc. 2006 Mar-Apr;13(2):121-6. doi: 10.1197/jamia.M2025. Epub 2005 Dec 15. PMID 16357345
- [Background] Jci. Joint Commission International Accreditation Standards for Hospitals. Jt Comm Resour Inc. 2013;5th Ed. doi:10.1017/CBO9781107415324.004.
- [Background] Tang PC, Black W, Young CY. Proposed criteria for reimbursing eVisits: content analysis of secure patient messages in a personal health record system. AMIA Annu Symp Proc. 2006;2006:764-8. PMID 17238444
- [Background] Tenforde M, Jain A, Hickner J. The value of personal health records for chronic disease management: what do we know? Fam Med. 2011 May;43(5):351-4. PMID 21557106
- [Background] Kaelber DC, Jha AK, Johnston D, Middleton B, Bates DW. A research agenda for personal health records (PHRs). J Am Med Inform Assoc. 2008 Nov-Dec;15(6):729-36. doi: 10.1197/jamia.M2547. Epub 2008 Aug 28. PMID 18756002
- [Background] Wells S, Rozenblum R, Park A, Dunn M, Bates DW. Organizational strategies for promoting patient and provider uptake of personal health records. J Am Med Inform Assoc. 2015 Jan;22(1):213-22. doi: 10.1136/amiajnl-2014-003055. Epub 2014 Oct 17. PMID 25326601
- [Background] Deterding S, Dixon D, Khaled R, Nacke L, Sicart M, O'Hara K. Gamification: Using Game Design Elements in Non-Game Contexts. Proc 2011 Annu Conf Ext Abstr Hum Factors Comput Syst (CHI 2011). 2011:2425-2428. doi:10.1145/1979742.1979575.
- [Background] Lister C, West JH, Cannon B, Sax T, Brodegard D. Just a fad? Gamification in health and fitness apps. JMIR Serious Games. 2014 Aug 4;2(2):e9. doi: 10.2196/games.3413. PMID 25654660
- [Background] King D, Greaves F, Exeter C, Darzi A. 'Gamification': influencing health behaviours with games. J R Soc Med. 2013 Mar;106(3):76-8. doi: 10.1177/0141076813480996. No abstract available. PMID 23481424
- [Background] McKeown S, Krause C, Shergill M, Siu A, Sweet D. Gamification as a strategy to engage and motivate clinicians to improve care. Healthc Manage Forum. 2016 Mar;29(2):67-73. doi: 10.1177/0840470415626528. Epub 2016 Feb 12. PMID 26872801
- [Background] Ryan RM, Deci EL. Self-determination theory and the facilitation of intrinsic motivation, social development, and well-being. Am Psychol. 2000 Jan;55(1):68-78. doi: 10.1037//0003-066x.55.1.68. PMID 11392867
- [Background] Mihaly Csikszentmihalyi. 1991. Flow: The psychology of optimal experience. HarperCollins Publishers, New York, New York, USA.